CLINICAL TRIAL: NCT03739060
Title: Impact of Transcutaneous Electric Nerve Stimulation (TENS) on Postoperative Pain and Quality of Life (QoL) After Inguinal Hernia Repair
Brief Title: Impact of TENS on Postoperative Pain and Quality of Life After Inguinal Hernia Repair
Acronym: TENS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Audrius Paršeliūnas, Principal Investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TENS1
Record Dates: First submitted 2018-10-23; First posted 2018-11-13 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Inguinal Hernia; Postoperative Pain; Quality of Life; Transcutaneous Electric Nerve Stimulation
Keywords: Inguinal hernia; Transcutaneous electric nerve stimulation; Postoperative pain; Quality of life; Pain threshold; Algometry
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TENS group (Active Comparator): Conventional transcutaneous electric nerve stimulation
  Interventions: Device: Transcutaneous electric nerve stimulation
- Placebo TENS group (Placebo Comparator): 0 amperes transcutaneous electric nerve stimulation
  Interventions: Device: Transcutaneous electric nerve stimulation

INTERVENTIONS:
Device: Transcutaneous electric nerve stimulation — Conventional transcutaneous electric nerve stimulation
  Other Names: TENS

SUMMARY:
Lichtenstein herniorrhaphy still remains one of the most often performed inguinal hernia repair techniques. It is frequently associated with acute postoperative and chronic pain. Due to insufficient effect of non-steroidal anti-inflammatory drugs, they are often overdosed. However opioids have many side effects. Interventional treatment, such as transversus abdominis plain (TAP) block requires an additional intervention and has relatively short effect, also could not be applied in outpatient conditions. The hypoalgesic effect of transcutaneous electric nerve stimulation (TENS) is well known for many years, but effectiveness during postoperative period is still controversial and maybe therefore didn't come to daily practice. However it could be a promising part of multi-modal pain treatment for hernia patients. This study analyse the hypoalgesic effect of TENS and its impact on hernia specific quality of life (QoL) after Lichtenstein hernia repair.

Aim#1 To determine whether use of TENS is effective for acute postoperative pain relief.

Aim#2 To determine whether use of TENS have impact on hernia specific QoL in early and late postoperative period.

Aim#3 To identify factors associated with effectiveness/ineffectiveness of TENS procedures.

Aim#4 To determine whether a psychological condition (depression, anxiety and pain catastrophisation) is somehow associated with TENS effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Elective Lichtenstein repair for primary hernia
* Male gender
* No TENS procedures in the past
* American Society of Anesthesiologists physical status I or II
* No cognitive, speaking, hearing or visual disturbances
* No movement disorders

Exclusion Criteria:

* Non Lithuanian speaker
* Known allergy to a patch glue
* Chronic use of non-steroidal anti inflammatory drugs or opioids
* Neuropathic diseases
* General contraindication for TENS procedures (such as skin disorders in site of electrodes application or pacemaker)
* Not able to complete the questionnaires

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-02-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Change in pain level as assessed by the VAS. | 10 min before and 10 min after each TENS procedure, which occur 24, 26, 48 and 50 hours after surgery.
  Pain is assessed using a 100 mm handheld slide rule-type visual analogue scale (VAS) with values from 0 to 100 (0 = no pain, 100 = extreme pain) during lying, waking and getting out of bed. Total scores are averaged.

SECONDARY OUTCOMES:
Change in pressure pain threshold. | 1 hour before surgery (baseline), 10 min before and 10 min after each TENS procedure, which occur 24, 26, 48 and 50 hours after surgery.
  Pressure pain threshold assessed using digital pressure algometer examination in inguinal region (hernia and contralateral side). Pressure in newtons (N) that evokes minimal sensation of pain is assessed.
Change in pressure pain tolerance. | 1 hour before surgery (baseline), 10 min before and 10 min after each TENS procedure, which occur 24, 26, 48 and 50 hours after surgery.
  Pressure pain tolerance assessed using digital pressure algometer examination in inguinal region (hernia and contralateral side). Pressure in newtons (N) that evokes maximal tolerable sensation of pain is assessed.
Change in hernia specific quality of life. | 1 hour before surgery (baseline), 2 days, 1 week, 4 weeks and 6 month after surgery.
  Hernia specific quality of life is assessed using self reported questionnaire Carolina's comfort scale (CCS) application, providing a 0 to 115 score.
Change in overall quality of life. | 1 hour before surgery (baseline), 2 days, 1 week, 4 weeks and 6 month after surgery.
  Overall quality of life is assessed using self reported short form (36) health survey questionnaire (SF-36) application.The SF-36 consists of 36 items, that aggregate into 8 parts: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Each domain is scored on a value of 0 (poor health) to 100 (best health).
Consumption of analgesic drugs. | 2 days postoperative
  The total amount of drugs, used for pain relief in hospital.
Depression status influence to TENS effectiveness. | 2 days postoperative
  Depression status is assessed using preoperative completed patient health questionnaire- 9 (PHQ-9), providing a 0 to 27 severity score.
Anxiety status influence to TENS effectiveness. | 2 days postoperative
  Anxiety status is assessed using preoperative completed generalized anxiety disorder scale -7 (GAD-7), providing a 0 to 21 severity score.
Pain catastrophizing influence to TENS effectiveness. | 2 days postoperative
  Pain catastrophizing is assessed using preoperative completed pain catastrophizing scale (PCS) questionnaire, providing a 0 to 52 score.

CONTACTS AND LOCATIONS:
Overall Officials: Audrius Paršeliūnas, MD, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

REFERENCES:
- [Derived] Parseliunas A, Paskauskas S, Kubiliute E, Vaitekunas J, Venskutonis D. Transcutaneous Electric Nerve Stimulation Reduces Acute Postoperative Pain and Analgesic Use After Open Inguinal Hernia Surgery: A Randomized, Double-Blind, Placebo-Controlled Trial. J Pain. 2021 May;22(5):533-544. doi: 10.1016/j.jpain.2020.11.006. Epub 2020 Dec 10. PMID 33309784